CLINICAL TRIAL: NCT03418155
Title: Efficacy and Safety of TongBi Capsule in Patients With Knee Osteoarthritis:a Randomized, Double-blind, Placebo-controlled Post - Market Clinical Study
Brief Title: Efficacy and Safety of TongBi Capsule in Patients With Knee Osteoarthritis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Quan Jiang, Director，Devision of Rheumatology, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BH_2016001
Record Dates: First submitted 2018-01-25; First posted 2018-02-01 (Actual); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment of TongBi Capsule (Experimental)
  Interventions: Drug: Treatment of TongBi Capsule
- Treatment of TongBi Placebo (Placebo Comparator)
  Interventions: Drug: Treatment of TongBi placebo

INTERVENTIONS:
Drug: Treatment of TongBi Capsule — TongBi Capsule:0.31g,3times a day, oral, for 4 weeks.
  Other Names: capsule A
  Arms: Treatment of TongBi Capsule
Drug: Treatment of TongBi placebo — TongBi placebo:0.31g,3times a day, oral, for 4 weeks.
  Arms: Treatment of TongBi Placebo

SUMMARY:
This study evaluates the efficacy and safety of TongBi capsule compared with placebo in the treatment of knee osteoarthritis in adults.Half of participants will receive TongBi capsule in combination,while the other half will receive a Placebo.

ELIGIBILITY:
Inclusion Criteria:

1.45-75 years of age (including 45 years and 75 years old), men and women are not limited.

2. western medicine diagnosis of knee osteoarthritis, clinical classification for primary.

3.The severity of the imaging classification of K-L≤Ⅲ; 4. treatment VAS pain scores than 40mm (select the subjects most obvious limb pain symptoms).

5. informed consent form signed by the patient or legal representative.

Exclusion Criteria:

1. within 3 months prior to the trial, the patients were treated within intra-articular treatment.
2. 4 weeks before the treatment, corticosteroids, non steroidal drugs, intra-articular injections or other drugs to improve the condition (such as cartilage protective agents) were used.
3. The screening period has any disease history or evidence:

   The basic of serious cardiovascular and cerebrovascular diseases; An active, recurrent peptic ulcer or other hemorrhagic disease risk; Sales and other serious diseases of digestive system; An associated with malignant tumors, blood, or other serious diseases or system; Patients who are unable to cooperate or cooperate with other mental disorders.
4. Before the screening, any laboratory test indicators meet the following standards:

   An admission of liver and kidney function showed that ALT and AST is more than 1.5 times the upper limit of the normal value, Cr is more than 1.2 times the upper limit of normal (Reference Research Center laboratory where the range of normal value); An other clinically significant laboratory abnormalities, and the researchers judged not into the group.
5. Allergic constitution or allergic to TongBi capsul, excipients or similar ingredients;
6. Professional athletes;
7. doubt or indeed history of alcohol and drug abuse;
8. participants who participated in other clinical trials within the first 3 months;
9. the researchers believe that patients should not participate in this clinical trial.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-02-01 (Estimated); Primary Completion 2019-04-01 (Estimated); Study Completion 2019-10-01 (Estimated)

PRIMARY OUTCOMES:
The change from Baseline to week 4 in Visual Analog Scale (VAS)score | 0 weeks,2 weeks，4 weeks
  VAS scores ranges from 0 to 100, with higher scores indicating heavier pain

SECONDARY OUTCOMES:
The change from Baseline to week 4 in Western Ontarioand McMaster Universities | 0 weeks,2 weeks and 4 weeks
  WOMAC scores ranges from 0 to 96, with higher scores indicating greater disability
The change from baseline to week 4 in The Short Form-36 Health Survey (SF-36) scores | 0 weeks,4 weeks
  SF-36 scores ranges from 0 to 100,it shows the extent of physical function
The number of adverse events | 4 weeks
  The number of adverse events related to treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jiang Quan, Principal Investigator — Guang'anmen Hospital of China Academy of Chinese Medical Sc
Locations (1):
- Guang'anmen Hospital of China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality, China